CLINICAL TRIAL: NCT06017583
Title: Neoadjuvant Chemotherapy With PD-1 Inhibitors Combined With Simultaneous Integrated Boost Intensity-modulated Radiotherapy in the Treatment of Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Chemotherapy With PD-1 Inhibitors Combined With SIB-IMRT in the Treatment of Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yong Zhang,MD (Other)
Responsible Party: Sponsor-Investigator, Yong Zhang,MD, First Affiliated Hospital of Guangxi Medical University, First Affiliated Hospital of Guangxi Medical University
Organization: First Affiliated Hospital of Guangxi Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-S845-01
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Rectal Neoplasms
Keywords: Rectal cancer; Tislelizumab; SIB IMRT
MeSH Terms: conditions — Rectal Neoplasms | interventions — tislelizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: The random number table method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): The experimental group will receive concurrent simultaneous integrated boost intensity-modulated radiotherapy (SIB-IMRT) and concurrent capecitabine chemotherapy, and complete 2 ~ 4 cycles of XELOX chemotherapy, while receiving full tislelizumab treatment for at least 4 cycles (21 days per cycle).
  Interventions: Drug: Tislelizumab; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: SIB-IMRT
- Control arm (Placebo Comparator): The control group received intensity-modulated radiotherapy (IMRT) without tirellizumab, and the other treatment regiments were consistent with the experimental group.
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Tislelizumab — Tirellizumab was administered intravenously at 200mg/d1, 21 days per cycle, with at least 4 cycles completed.
  Arms: Experimental arm
Drug: Capecitabine — Oral capecitabine 825mg/m2 bid, radiotherapy day concurrent chemotherapy. Chemotherapy regimen after radiotherapy: XELOX regimen: oxaliplatin intravenous infusion of 130mg/m2/d1+ oral capecitabine 1000mg/m2 bid/ d1-14, 21 days per cycle, at least 2 cycles completed.
Drug: Oxaliplatin — Chemotherapy regimen after radiotherapy: XELOX regimen: oxaliplatin intravenous infusion of 130mg/m2/d1+ oral capecitabine 1000mg/m2 bid/ d1-14, 21 days per cycle, at least 2 cycles completed.
Radiation: SIB-IMRT — The tumor and the related mesenteric region 1cm above and below were simultaneously integrated boost to 5600cGy with the intensity-modulated radiotherapy. The other dose for clinical target volume is 5000 cGy.
  Arms: Experimental arm
Radiation: IMRT — The whole dose of the clinical target volume is 5000 cGy with intensity-modulated radiotherapy.
  Arms: Control arm

SUMMARY:
This study aims to evaluate the efficacy and safety of tislelizumab combined with simultaneous integrated boost intensity-modulated radiotherapy in treating locally advanced rectal cancer. To explore a new PD-1 inhibitor adjuvant chemotherapy model combined with radiotherapy to treat locally advanced rectal cancer.

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT). Patients with T3-4 in the 8th AJCC stage or positive regional lymph nodes and no distant metastases will be enrolled. Forty-eight patients will be enrolled by inclusion and exclusion criteria. The enrolled patients will be randomly divided into experimental and control groups (twenty-four patients for each group) to receive preoperative neoadjuvant therapy. The experimental group will receive concurrent simultaneous integrated boost intensity-modulated radiotherapy (SIB-IMRT) and concurrent capecitabine chemotherapy, and complete 2 ~ 4 cycles of XELOX chemotherapy, while receiving complete tislelizumab treatment for at least 4 cycles (21 days per cycle). The control group received intensity-modulated radiotherapy (IMRT) without tirellizumab, and the other treatment regiments were consistent with the experimental group. The tumor size will be measured in MRI or CT images, and side effects will be recorded. The primary outcome was CR rate (pathological complete response rate and clinical complete response rate), and secondary outcomes were side effects and 3-year OS and DFS.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years.
2. The pathological type of rectal cancer diagnosed by histopathology is adenocarcinoma.
3. Patients with T3-4 in the eighth AJCC stage or positive regional lymph node and no distant metastasis.
4. Having at least one measurable lesion according to RECIST 1.1.
5. ECOG score 0-1.
6. Expected survival time ≥6 months.
7. Major organ function is normal, that is, meeting the following criteria: blood routine: HB≥90g/L, ANC≥1.5×109/L, PLT≥80×109/L; Biochemical examination of ALB≥30g/L, TBIL≤1.5 ULN, ALT and AST≤2.5 ULN, plasma Cr≤1.5 ULN or creatinine clearance ≥60 ml/min.
8. Subjects volunteered to join the study, signed the informed consent, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Patients have had or currently have other malignant tumors within 5 years.
2. Patients allergic or sensitive to any drug in the study protocol.
3. Patients innate or acquired immune deficiency (e.g. HIV infection).
4. The presence of any active, known or suspected autoimmune disease (such as, but not limited to, interstitial pneumonia, uveitis, enteritis, hepatitis, arthritis, nephritis, hypophysitis, hyperthyroidism, hypothyroidism, etc.); The subject had vitiligo. Subjects with asthma require bronchodilators for medical intervention.
5. The presence of active infections requiring systemic treatment.
6. The subject has previously received other PD-1 or PD-L1, or CTLA-4 antibody therapy, or other drug therapy targeting immunoregulatory receptor preparations.
7. Unrelieved toxic effects above CTCAE grade 1 due to any previous treatment, excluding alopecia.
8. Patients with a history of myocardial infarction or stroke, unstable angina pectoris, decompensated heart failure or deep vein thrombosis.
9. Patients with long-term untreated wounds or fractures, major surgical operations or severe traumatic injuries, fractures or ulcers within 4 weeks.
10. Pregnant or lactating women.
11. Patients with liver and kidney dysfunction.
12. Patients with a history of abuse of psychotropic drugs and unable to abstain or patients with mental disorders.
13. Patients who have participated in clinical trials of other drugs within 4 weeks.
14. Patients with concomitant diseases that, in the judgment of the investigator, seriously endanger the patient's safety or affect the patient's completion of the study.
15. The investigator judged that participation in this study was not conducive to the maximum benefit of the subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 12 weeks~18 weeks
  Include in pathological complete response rate and clinical complete response rate. MRI/CT will be used for evaluating the carcinoma status. Pathological complete response rate will be evaluated by surgery.

SECONDARY OUTCOMES:
Side effects | 6monthes, 3years
  Myelosuppression, radiation enteritis, radiothermitis
Overall survival | 3 years
  OS was calculated from the date of entry into the study to the date of death or the last follow-up visit.
Disease free survival | 3 years
  DFS was calculated from the date of entry into the study to the date of the time from the beginning of randomization to the disease recurrence or progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No